CLINICAL TRIAL: NCT03022292
Title: The IAI-OCTA Study or; Microvascular Structure and Morphology of Neovascular Membranes in Age Related Macular Degeneration (AMD) After Intravitreal Aflibercept Injection (IAI) Therapy Using OCT-Angiography Analysis
Brief Title: The IAI-OCTA Study; a Study of OCT-Angiography Analysis Efficacy
Acronym: IAI-OCTA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, David Sarraf, MD, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16-000925
Record Dates: First submitted 2016-11-10; First posted 2017-01-16 (Estimated); Results first posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Wet Macular Degeneration
MeSH Terms: conditions — Wet Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- IAI Treatment (Experimental): Intravitreal injection of aflibercept 2 mg/0.05 ml at baseline, week 4, week 8, week 16, week 24, week 36, and week 48. Additional injections can be administered during the remaining visits on an as needed basis per Primary Investigator (PI) discretion based on the presence of any intraretinal or subretinal fluid on OCT, heme visualized on examination, reduction of BCVA by 5 or more ETDRS letters, or evidence of either increased area, density, or activity of the brush border of the neovascularization on OCT-angiography. There will be a minimum of 21 days between subsequent injections. Each subject will therefore receive a minimum of 7 injections and up to a maximum of 13 injections throughout the study period.
  Interventions: Drug: Aflibercept Ophthalmic; Device: optovue angiovue

INTERVENTIONS:
Drug: Aflibercept Ophthalmic — IAI given for active exudative macular degeneration (CNV, SRF, PED) per SOC
Device: optovue angiovue — FDA approved Optovue Angiovue will be used to monitor progression and responsiveness of active exudative macular degeneration to IAI.
  Other Names: OCTA

SUMMARY:
A study investigating the ability of OCTA imaging technology to identify and analyze untreated type 1, 2, and 3 neovascular membrane lesions in treatment naive patients with exudative macular degeneration, as well as investigating the ability of the OCTA imaging technology to evaluate the treatment outcomes of Intravitreal Aflibercept Injection in neovascular lesions associated with macular degeneration.

This study is utilizing a new, FDA approved, non-standard of care technology (OCT-Angiography by Optovue) to image and evaluate the treatment outcomes of using standard of care Intravitreal Aflibercept Injections for their approved use in patients diagnosed with neovascular AMD who are naive to previous Anti-VEGF therapies.

DETAILED DESCRIPTION:
Prospective study of neovascular AMD subjects with type 1, 2, or 3 neovascularization that have not been treated with prior anti-VEGF therapy. Subjects will be scheduled for intravitreal aflibercept injection (IAI) at baseline, week 4, week 8, week 16, week 24, week 36, and week 48. Additional injections can be administered during the remaining visits on an as needed basis per PI discretion based on the presence of any intraretinal or subretinal fluid on OCT, heme visualized on examination, reduction of BCVA by 5 or more ETDRS letters, or evidence of either increased area, density, or activity of the brush border of the neovascularization on OCT angiography. There will be a minimum of 21 days between subsequent injections. Each subject will therefore receive a minimum of 7 injections and up to a maximum of 13 injections throughout the study period. No injection will be given on the exit visit, week 52. OCT angiography and spectral domain OCT imaging will be performed at baseline and every 4 weeks thereafter

The above procedures are standard of care for neovascular AMD subjects.

As part of this study, these subjects will also undergo imaging of both eyes with OCTA at each visit. This is not standard of Care and is research.

The only procedure that is being performed for research is the OCT-A. The injections and all other procedure are SOC based on physician discretion and clinical need. The investigators will not be modifying the dosage amounts or frequency.

A subgroup of willing subjects will undergo OCT angiography every 2 weeks for the first 12 weeks.

Indocyanine green angiography will be performed at baseline for all subjects to establish baseline subject population characteristics. Fluorescein angiography will be performed at baseline, week 12, and week 52 for efficacy monitoring. Detailed OCT angiography analysis will be performed to identify anatomical and morphological biomarkers of growth progression and disease activity. In addition to qualitative structural and morphological analysis, detailed quantitative OCT angiography analysis of the neovascular lesion using automated or manual capillary density maps and area calculation will be performed at each visit to determine the detailed microvascular response of neovascular complexes to IAI therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is older than 50 years of age.
2. Subject is willing to participate in the study and able to follow the study criteria and protocol.
3. The study eye is treatment naive regarding treatment of neovascular AMD.
4. Subject is willing and able to comply with clinic visits and study-related procedures.
5. Subject is able to provide signed informed consent.
6. Subject is able to understand and complete study-related questionnaires.
7. The subject is not currently involved with any other clinical study.
8. Best Corrected Visual Acuity (BCVA) with ETDRS Snellen equivalent of 20/400 or better and 20/32 or worse.
9. Sufficiently clear media (cornea, anterior chamber, lens, vitreous) for OCT, FA and fundus photography (FP).
10. Intraocular pressure (IOP) of 25mmHg or less in the study eye, with or without use of ocular hypotensive agents.
11. Prior focal corticosteroid treatment is allowed, as long as the study eye is not involved. However prior (within 90 days of Day 0) or current systemic corticosteroid therapy (oral or intravenous corticosteroid treatment) is not permitted.

Exclusion Criteria:

1. Any prior treatment of neovascular AMD in the eye proposed for enrollment including previous anti-vascular endothelial factor (anti-VEGF) therapy, photodynamic therapy (PDT), radiation therapy, corticosteroid treatment, surgical treatment for CNV, thermal laser treatment, and any other prior intravitreal treatment for neovascular AMD (except minerals and vitamins).
2. Known serious allergies to aflibercept, fluorescein dye, Indocyanine Green (ICG), shellfish, drugs for pupillary dilation, topical anesthetic, or sterilizing solution (e.g. Betadine Solution).
3. Prior or current systemic anti-VEGF therapy.
4. Pregnant or breast-feeding women.
5. Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly).
6. Contraindication to pupillary dilation in study eye.
7. Any condition (including inability to read visual acuity charts, or language barrier) that may preclude subjects ability to comply with the study protocol and requirements.
8. Presence of any advanced systemic condition or end-stage disease, such as advanced Alzheimer Syndrome, end-stage cancer, etc., which will likely prevent subject from completing study.
9. Previous therapeutic radiation in the region of the study eye.
10. Prior retinal pigment epithelial (RPE) tear in study eye.
11. Prior ocular surgery (except YAG laser capsulotomy) for study within the past 90 days.
12. Anticipated ocular surgery (except YAG laser capsulotomy) for the next 12 months.
13. Prior vitrectomy in the study eye.
14. Presence of any causes of CNV and PED other than due to AMD or presence of ocular disease other than AMD affecting study eye, i.e. presumed ocular histoplasmosis syndrome, android streaks, pathologic myopia

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stein Eye Institute of UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Congdon N, O'Colmain B, Klaver CC, Klein R, Munoz B, Friedman DS, Kempen J, Taylor HR, Mitchell P; Eye Diseases Prevalence Research Group. Causes and prevalence of visual impairment among adults in the United States. Arch Ophthalmol. 2004 Apr;122(4):477-85. doi: 10.1001/archopht.122.4.477. PMID 15078664
- [Background] Solomon SD, Lindsley K, Vedula SS, Krzystolik MG, Hawkins BS. Anti-vascular endothelial growth factor for neovascular age-related macular degeneration. Cochrane Database Syst Rev. 2014 Aug 29;8(8):CD005139. doi: 10.1002/14651858.CD005139.pub3. PMID 25170575
- [Background] Kuehlewein L, Bansal M, Lenis TL, Iafe NA, Sadda SR, Bonini Filho MA, De Carlo TE, Waheed NK, Duker JS, Sarraf D. Optical Coherence Tomography Angiography of Type 1 Neovascularization in Age-Related Macular Degeneration. Am J Ophthalmol. 2015 Oct;160(4):739-48.e2. doi: 10.1016/j.ajo.2015.06.030. Epub 2015 Jul 9. PMID 26164826
- [Background] Kuehlewein L, Dansingani KK, de Carlo TE, Bonini Filho MA, Iafe NA, Lenis TL, Freund KB, Waheed NK, Duker JS, Sadda SR, Sarraf D. OPTICAL COHERENCE TOMOGRAPHY ANGIOGRAPHY OF TYPE 3 NEOVASCULARIZATION SECONDARY TO AGE-RELATED MACULAR DEGENERATION. Retina. 2015 Nov;35(11):2229-35. doi: 10.1097/IAE.0000000000000835. PMID 26502007
- [Background] Miere A, Querques G, Semoun O, El Ameen A, Capuano V, Souied EH. OPTICAL COHERENCE TOMOGRAPHY ANGIOGRAPHY IN EARLY TYPE 3 NEOVASCULARIZATION. Retina. 2015 Nov;35(11):2236-41. doi: 10.1097/IAE.0000000000000834. PMID 26457399
- [Background] El Ameen A, Cohen SY, Semoun O, Miere A, Srour M, Quaranta-El Maftouhi M, Oubraham H, Blanco-Garavito R, Querques G, Souied EH. TYPE 2 NEOVASCULARIZATION SECONDARY TO AGE-RELATED MACULAR DEGENERATION IMAGED BY OPTICAL COHERENCE TOMOGRAPHY ANGIOGRAPHY. Retina. 2015 Nov;35(11):2212-8. doi: 10.1097/IAE.0000000000000773. PMID 26441269
- [Background] Jia Y, Bailey ST, Wilson DJ, Tan O, Klein ML, Flaxel CJ, Potsaid B, Liu JJ, Lu CD, Kraus MF, Fujimoto JG, Huang D. Quantitative optical coherence tomography angiography of choroidal neovascularization in age-related macular degeneration. Ophthalmology. 2014 Jul;121(7):1435-44. doi: 10.1016/j.ophtha.2014.01.034. Epub 2014 Mar 27. PMID 24679442
- [Background] Miere A, Semoun O, Cohen SY, El Ameen A, Srour M, Jung C, Oubraham H, Querques G, Souied EH. OPTICAL COHERENCE TOMOGRAPHY ANGIOGRAPHY FEATURES OF SUBRETINAL FIBROSIS IN AGE-RELATED MACULAR DEGENERATION. Retina. 2015 Nov;35(11):2275-84. doi: 10.1097/IAE.0000000000000819. PMID 26457397
- [Background] Coscas G, Lupidi M, Coscas F, Francais C, Cagini C, Souied EH. Optical coherence tomography angiography during follow-up: qualitative and quantitative analysis of mixed type I and II choroidal neovascularization after vascular endothelial growth factor trap therapy. Ophthalmic Res. 2015;54(2):57-63. doi: 10.1159/000433547. Epub 2015 Jul 17. PMID 26201877
- [Background] Spaide RF. Optical Coherence Tomography Angiography Signs of Vascular Abnormalization With Antiangiogenic Therapy for Choroidal Neovascularization. Am J Ophthalmol. 2015 Jul;160(1):6-16. doi: 10.1016/j.ajo.2015.04.012. Epub 2015 Apr 14. PMID 25887628
- [Background] Schmidt-Erfurth U, Kaiser PK, Korobelnik JF, Brown DM, Chong V, Nguyen QD, Ho AC, Ogura Y, Simader C, Jaffe GJ, Slakter JS, Yancopoulos GD, Stahl N, Vitti R, Berliner AJ, Soo Y, Anderesi M, Sowade O, Zeitz O, Norenberg C, Sandbrink R, Heier JS. Intravitreal aflibercept injection for neovascular age-related macular degeneration: ninety-six-week results of the VIEW studies. Ophthalmology. 2014 Jan;121(1):193-201. doi: 10.1016/j.ophtha.2013.08.011. Epub 2013 Sep 29. PMID 24084500

RESULTS

PARTICIPANT FLOW:
Groups:
- IAI Treatment: Intravitreal injection of aflibercept 2 mg/0.05 ml at baseline, week 4, week 8, week 16, week 24, week 36, and week 48.
  Aflibercept Ophthalmic: IAI given for active exudative macular degeneration (CNV, SRF, PED) per SOC
  optovue angiovue: FDA approved Optovue Angiovue will be used to monitor progression and responsiveness of active exudative macular degeneration to IAI.
Period: Overall Study
Arm/Group | IAI Treatment
Started | 26
Completed | 24
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | IAI Treatment
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 19
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 26
Mean BCVA in LogMAR [Mean (Full Range); unit: score] — Best Corrected Visual acuity (BCVA) was assessed at a distance of 4 meters from Snellen and converted to logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with a lower logMAR value indicating better visual acuity. Population: Measure includes all participants with analyzable baseline BCVA
  score
    number analyzed (Participants) | 25
    (all) | 0.32 [-0.2 to 1.3]
OCTA Analysis of Lesion Area [Mean (Full Range); unit: mm^2] | 2.008 [0 to 18.016]

OUTCOME MEASURES:

1. Primary Outcome: Area of Lesion Measured by Optical Coherence Tomography Angiography (OCTA) Scan.
Description: Area of the neovascular lesion (in millimeters^2)
Time Frame: Week 24
Population: Participants present for 24 week assessment
Measure: Mean (Full Range); unit: mm^2
Arm/Group | IAI Treatment
Number analyzed (Participants) | 24
mm^2 | 1.07 [0 to 9.939]

2. Primary Outcome: Area of Lesion Measured by Optical Coherence Tomography Angiography (OCTA) Scan.
Description: Area of the neovascular lesion (in millimeters^2)
Time Frame: Week 52
Population: Participants present for 52 week assessment
Measure: Mean (Full Range); unit: mm^2
Arm/Group | IAI Treatment
Number analyzed (Participants) | 20
mm^2 | 0.67 [0 to 6.056]

3. Secondary Outcome: Best Corrected Visual Acuity (BCVA) -Early Treatment Diabetic Retinopathy Study (ETDRS) Letter Change
Description: patients with gain of ≥5, ≥10, or ≥15 ETDRS letters. The ETDRS chart is read at 4.0 meters, and presents a series of five letters of equal difficulty on each row, with standardized spacing between letters and rows, for a total of 14 lines (70 letters).
Time Frame: Baseline, Week 24
Population: Participants with analyzable ETDRS at both baseline & week 24
Measure: Number; unit: participants
Arm/Group | IAI Treatment
Number analyzed (Participants) | 23
participants
  ≥5 ETDRS letters | 4
  ≥10 ETDRS letters | 2
  ≥15 ETDRS letters | 0

4. Secondary Outcome: Best Corrected Visual Acuity (BCVA) -ETDRS Letter Change
Description: as for outcome 3
Time Frame: Week 24, Week 52
Population: Participants with analyzable BCVA at both 24 and 52 weeks
Measure: Number; unit: participants
Arm/Group | IAI Treatment
Number analyzed (Participants) | 21
participants
  ≥5 ETDRS letters | 4
  ≥10 ETDRS letters | 1
  ≥15 ETDRS letters | 0

5. Secondary Outcome: Mean Best Corrected Visual Acuity (BCVA)
Description: Visual acuity (VA) was assessed at a distance of 4 meters from Snellen and converted to logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with a lower logMAR value indicating better visual acuity.
Time Frame: Week 24
Population: Participants with analyzable measure at week 24
Measure: Mean (Full Range); unit: score
Arm/Group | IAI Treatment
Number analyzed (Participants) | 24
score | 0.3 [-0.2 to 1.3]

6. Secondary Outcome: Mean Best Corrected Visual Acuity (BCVA)
Description: as for outcome 5
Time Frame: Week 52
Population: Participants with analyzable BCVA at 52 weeks
Measure: Mean (Full Range); unit: score
Arm/Group | IAI Treatment
Number analyzed (Participants) | 22
score | 0.33 [-0.2 to 1.2]

7. Other Pre Specified Outcome: OCTA Neovascular Membrane Regression Ratio of Change
Description: OCT angiography regression of neovascular membrane as measured by ratio of change in area of the neovascular lesion (in millimeters^2) during the initial 12 weeks
Time Frame: 12 weeks
Measure: Mean (Inter-Quartile Range); unit: ratio
Arm/Group | IAI Treatment
Number analyzed (Participants) | 26
ratio | 0.37 [0.14 to 0.74]

8. Other Pre Specified Outcome: Presence of Intraretinal and Subretinal Fluid, and Subretinal Hyper-Reflective Material (SHRM) on Spectral Domain Optical Coherence Tomography (SD-OCT) Scan.
Description: Participants with presence of intraretinal and subretinal fluid, and Subretinal Hyper-Reflective Material (SHRM)
Time Frame: week 24
Population: Participants present for assessment at week 24
Measure: Count of Participants; unit: Participants
Arm/Group | IAI Treatment
Number analyzed (Participants) | 24
Participants
  intraretinal | 4
  subretinal | 9
  SHRM | 1

9. Other Pre Specified Outcome: SD OCT Presence of Intraretinal and Subretinal Fluid, and Subretinal Hyper-Reflective Material (SHRM)
Description: Participants with presence of SD OCT intraretinal and subretinal fluid, and Subretinal Hyper-Reflective Material (SHRM)
Time Frame: week 52
Population: Participants present for assessment at 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | IAI Treatment
Number analyzed (Participants) | 22
Participants
  intraretinal | 3
  subretinal | 6
  SHRM | 0

10. Other Pre Specified Outcome: Ocular AE
Description: ocular adverse events
Time Frame: 52 weeks
Population: All participants at risk for AE
Measure: Number; unit: events
Arm/Group | IAI Treatment
Number analyzed (Participants) | 26
events | 2

11. Other Pre Specified Outcome: Relevant Systemic SAE
Description: relevant systemic serious adverse events
Time Frame: 52 weeks
Population: Participants at risk for AE during study
Measure: Number; unit: events
Arm/Group | IAI Treatment
Number analyzed (Participants) | 26
events | 1

12. Other Pre Specified Outcome: Number of Injections
Time Frame: week 24
Population: Participants present at week 24 visit
Measure: Number; unit: injections
Arm/Group | IAI Treatment
Number analyzed (Participants) | 25
injections | 25

13. Other Pre Specified Outcome: Number of Injections
Time Frame: week 52
Population: Participants present for week 52 visit
Measure: Number; unit: injections
Arm/Group | IAI Treatment
Number analyzed (Participants) | 22
injections | 12

14. Other Pre Specified Outcome: OCTA Neovascular Membrane Biomarker Qualitative Analysis (Sub-study)
Description: In subjects participating in the sub-study of serial OCT Angiography during the initial 12 weeks OCT angiography qualitative analysis of morphological biomarkers of the neovascular complex including attenuation of the fringe during the initial 12 weeks
Time Frame: Week 1-12
Population: Qualitative analyses not performed due to study staff turnover and lack of expertise
Arm/Group | IAI Treatment
Number analyzed (Participants) | 0

15. Other Pre Specified Outcome: SD OCT Analysis of Central Macular Thickness
Description: Ratio of change in SD OCT central macular thickness, calculated as change between visits divided by baseline measure.
Time Frame: Baseline to week 24
Population: Participants present for both baseline and week 24 assessment
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | IAI Treatment
Number analyzed (Participants) | 24
ratio | 0.08 (0.27)

16. Other Pre Specified Outcome: SD OCT Analysis of Central Macular Thickness
Description: Ratio of change in SD OCT central macular thickness, calculated as change between visits divided by baseline measure.
Time Frame: Baseline to week 52
Population: Participants present for both baseline and week 52 assessment
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | IAI Treatment
Number analyzed (Participants) | 24
ratio | 0.07 (0.25)

17. Other Pre Specified Outcome: OCTA Analysis of Vessel Density
Description: OCT angiography ratio of change in neovascular membrane as measured by area of the neovascular lesion in mm^2 at baseline and week 24. Ratio of change was calculated as change from baseline divided by the baseline value.
Time Frame: 24 weeks
Population: Participants present for both baseline and 24 week assessment
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | IAI Treatment
Number analyzed (Participants) | 24
ratio | -0.12 (2.73)

18. Other Pre Specified Outcome: OCTA Neovascular Membrane Biomarker Qualitative Analysis of Flow-void Areas(Sub-study)
Description: In subjects participating in the sub-study of serial OCT Angiography during the initial 12 weeks) OCT angiography qualitative analysis of morphological biomarkers of the neovascular complex including presence of flow-void areas during the initial 12 weeks
Time Frame: Week 1-12
Population: Qualitative analyses not performed due to study staff turnover and lack of expertise
Arm/Group | IAI Treatment
Number analyzed (Participants) | 0

19. Other Pre Specified Outcome: OCTA Neovascular Membrane Biomarker Qualitative Analysis of Vessel Looping (Sub-study)
Description: In subjects participating in the sub-study of serial OCT Angiography during the initial 12 weeks) OCT angiography qualitative analysis of morphological biomarkers of the neovascular complex including changes in vessel looping during the initial 12 weeks
Time Frame: Week 1-12
Population: Qualitative analyses not performed due to study staff turnover and lack of expertise
Arm/Group | IAI Treatment
Number analyzed (Participants) | 0

20. Other Pre Specified Outcome: SD OCT Analysis of SRF Volume
Description: Change in volume of subretinal fluid
Time Frame: week 24 and 52
Population: Fluid volume measures not performed due to study staff turnover and lack of expertise
Arm/Group | IAI Treatment
Number analyzed (Participants) | 0

21. Other Pre Specified Outcome: SD OCT Analysis of SHRM Volume
Description: Change volume of SHRM
Time Frame: week 24 and 52
Population: Fluid volume measures not performed due to study staff turnover and lack of expertise
Arm/Group | IAI Treatment
Number analyzed (Participants) | 0

22. Other Pre Specified Outcome: Presence of CME (Cystoid Macular Edema) on Spectral Domain Optical Coherence Tomography (SD-OCT) Scan.
Description: Participants with presence of cystoid macular edema
Time Frame: week 24
Population: Participants assessed for CME at week 24
Measure: Count of Participants; unit: Participants
Arm/Group | IAI Treatment
Number analyzed (Participants) | 23
Participants | 4

23. Other Pre Specified Outcome: Presence of CME (Cystoid Macular Edema) on Spectral Domain Optical Coherence Tomography (SD-OCT) Scan.
Description: Participants with presence of cystoid macular edema
Time Frame: week 52
Population: Participants assessed for CME at week 52
Measure: Count of Participants; unit: Participants
Arm/Group | IAI Treatment
Number analyzed (Participants) | 23
Participants | 3

24. Other Pre Specified Outcome: Pigment Epithelial Detachment (PED) Volume as Determined by SD OCT Analysis
Description: Change in ratio of volume of pigment epithelial detachment (PED), calculated as change from baseline divided by baseline value.
Time Frame: Baseline to week 24
Population: Participants present for both baseline and week 24 assessment
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | IAI Treatment
Number analyzed (Participants) | 24
ratio | 0.18 (0.6)

25. Other Pre Specified Outcome: PED Volume as Determined by SD OCT Analysis
Description: Change in ratio of volume of PED, calculated as change from baseline divided by baseline value.
Time Frame: Baseline to Week 52
Population: Participants present for both baseline and week 52 assessment
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | IAI Treatment
Number analyzed (Participants) | 24
ratio | 0.08 (0.9)

26. Other Pre Specified Outcome: PED Height as Determined by SD OCT Analysis
Description: Ratio of change in height of PED, calculated as change from baseline divided by baseline value
Time Frame: Baseline, week 24
Population: Participants present for both baseline and week 24 assessment
Measure: Mean (Inter-Quartile Range); unit: ratio
Arm/Group | IAI Treatment
Number analyzed (Participants) | 24
ratio | 0.26 [0.03 to 0.51]

27. Other Pre Specified Outcome: PED Height as Determined by SD OCT Analysis
Description: Ratio of change in height of PED, calculated as change from baseline divided by baseline value
Time Frame: Baseline, week 52
Population: Participants present for both baseline and week 52 assessment
Measure: Mean (Inter-Quartile Range); unit: ratio
Arm/Group | IAI Treatment
Number analyzed (Participants) | 24
ratio | 0.38 [0.12 to 0.67]

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | IAI Treatment
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 1/26
Other Adverse Events (participants affected / at risk) | 2/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IAI Treatment (N=26)
Retinal detachment (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IAI Treatment (N=26)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/92/NCT03022292/Prot_SAP_000.pdf